CLINICAL TRIAL: NCT00842140
Title: Metabolic Effects of Multiple Therapies in Polycystic Ovary Syndrome (PCOS) Women
Brief Title: Safety of Hormonal Contraceptives Therapies in Polycystic Ovary Syndrome (PCOS) Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Rui Alberto Ferriani, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRP15811/2005
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2009-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; Oral Contraceptives, Hormonal; Cardiovascular Disease; Endothelium
MeSH Terms: conditions — Polycystic Ovary Syndrome; Cardiovascular Diseases | interventions — Contraceptives, Oral; Belara; Spironolactone; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): This group will receive an oral contraceptive containing 0,03mg ethynylestradiol and 2mg chlormadinone acetate
  Interventions: Drug: oral contraceptive
- 2 (Experimental): The patient will receive an oral contraceptive (0,03mg ethynylestradiol and 2mg chlormadinone acetate) plus 100 mg spironolactone. One pill each once a day for twelve months.
  Interventions: Drug: Oral contraceptive plus spironolactone
- 3 (Experimental): The patient will receive an oral contraceptive (0,03mg ethynylestradiol and 2mg chlormadinone acetate) plus 850 mg metformin.
  Interventions: Drug: Oral contraceptive plus metformin

INTERVENTIONS:
Drug: oral contraceptive — oral contraceptive (0,03mg ethynylestradiol and 2mg chlormadinone acetate)once a day for 12 months
  Other Names: Belara
  Arms: 1
Drug: Oral contraceptive plus spironolactone — The patient will receive an oral contraceptive (0,03mg ethynylestradiol and 2mg chlormadinone acetate) plus 100 mg spironolactone. One pill each once a day for twelve months.
  Other Names: Belara; Spironolactone
  Arms: 2
Drug: Oral contraceptive plus metformin — Oral contraceptive (0,03mg ethynylestradiol and 2mg chlormadinone acetate) plus 850 mg of metformin
  Other Names: Belara; Metformin
  Arms: 3

SUMMARY:
The purpose of this study to assess early markers of cardiovascular disease in women with polycystic ovary syndrome in use of oral contraceptive containing ethynilestradiol and chlormadinone acetate alone or associated with Spironolactone.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is associated with comorbidities that may contribute to increased risk of cardiovascular disease (CVD). Oral contraceptives (OC) have been the mainstay of PCOS pharmacological therapy for decades. However, in non-hyperandrogenic women, OC use is associated with higher risk of cardiovascular disease, raising concern about a possible worsening of the unfavorable metabolic and cardiovascular profile of PCOS patients. There is lack of evidence about the impact of PCOS pharmacological therapies on cardiovascular risk markers and the long-term safety of these drugs in PCOS has not been established. The aim of this study is to compare the effect of an OC alone or associated with an anti-androgenic drug (spironolactone) on echografic cardiovascular risk markers, metabolic and hemostatic variables.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 35 years
* diagnosis of PCOS by Rotterdam Consensus

Exclusion Criteria:

* smoking, alcoholism, drug addiction;
* current pregnancy;
* current or previous use (up to two months before the study) of oral, vaginal, monthly injectable, or transdermal combined hormonal contraceptives;
* current or previous use (up to six months before the study) of a long-lasting hormonal contraceptive method (injectable, implant, or intrauterine device);
* antiandrogenic or hypoglycemic drugs, anti-inflammatory drugs, or statins;
* presence of systemic diseases (DM2, cardiovascular disease, autoimmune diseases, liver disease, thyroid disease, or congenital renal hyperplasia);
* personal history of arterial or venous thrombosis; chronic or acute inflammatory processes;
* puerperium of 12 weeks or less

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2006-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To compare the effect of an oral contraceptive alone or associated with an anti-androgenic drug (spironolactone) or associated with metformin on echografic cardiovascular risk markers. | 12 months

SECONDARY OUTCOMES:
to compare the effect of an oral contraceptive alone or associated with an anti-androgenic drug (spironolactone) or associated with metformin on seric cardiovascular risk markers. | 12 months
to compare the effect of an oral contraceptive alone or associated with an anti-androgenic drug (spironolactone) or associated with metformin on hemostatic variables. | 12 months
to compare the effect of an oral contraceptive alone or associated with an anti-androgenic drug (spironolactone) or associated with metformin on metabolic variables. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rui A Ferriani, MD, PhD, Study Director — University of Sao Paulo; Marcos Felipe S de Sa, MD, PhD, Study Chair — University of Sao Paulo; Carolina S Vieira, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil